CLINICAL TRIAL: NCT01342120
Title: Seroquel Safety Study
Brief Title: PHARMO Institute Seroquel Safety Study
Acronym: PHARMO II
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: PHARMO Institute for Drug Outcomes Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: D1443L00085
Record Dates: First submitted 2011-04-21; First posted 2011-04-27 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Schizophrenia; Major Depressive Disorder; Bipolar Disorder; Generalized Anxiety Disorder
Keywords: atypical antipsychotics; quetiapine
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major; Bipolar Disorder; Generalized Anxiety Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Quetiapine: Quetipine users
- All other atypical antipsychotics: All other atypical antipsychotics users
- Risperidone: Risperidone users
- Olanzapine: Olanzapine users

SUMMARY:
The purpose of this observational study is to study specific outcomes of interest in users of quetiapine compared with all other atypical antipsychotics and specifically olanzapine and risperidone. The outcomes of interest are all-cause mortality, failed suicide attempts, extrapyramidal symptoms, diabetes mellitus, hypothyroidism, acute myocardial infarction and stroke. This retrospective cohort study is based on population-based record linkage system (PHARMO RLS) capturing about 2.5 millions residents in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Episode of new use of atypical antipsychotics in naïve (not used antipsychotic drugs for a year) users of antipsychotics.

Exclusion Criteria:

* less than a year of recorded history before the cohort entry date
* use of multiple antipsychotics concomitantly
* duration and dose of the antipsychotic drug cannot be determined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population based sample of about 2.5 millions residents in the Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 18325 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The outcomes of interest will be evaluated by means of relative risk based on incidence rates estimates in users of quetiapine vs corresponding incidence rates in users of comparison drugs

CONTACTS AND LOCATIONS:
Overall Officials: Edith Heintjes, Principal Investigator — PHARMO Institute for Drug Outcomes Research

REFERENCES:
- [Derived] Heintjes EM, Overbeek JA, Penning-van Beest FJ, Brobert G, Herings RM. Post authorization safety study comparing quetiapine to risperidone and olanzapine. Hum Psychopharmacol. 2016 Jul;31(4):304-12. doi: 10.1002/hup.2539. Epub 2016 Jun 13. PMID 27297785